CLINICAL TRIAL: NCT06716255
Title: Observational Single-center Comparative Study of the Efficacy of Buffered Acetylsalicylic Acid and Enteric-coated Acetylsalicylic Acid on Platelet Aggregation in Patients With Chronic Coronary Syndrome and Type 2 Diabetes Mellitus
Brief Title: Comparison of Effects of Buffered and Enteric-coated Forms of Aspirin on Platelet Aggregation in Patients With Diabetes Mellitus and Chronic Coronary Syndrome
Acronym: CASCADE
Status: Completed | Type: Observational
Sponsor: Nizhpharm (Other)
Collaborators: Federal Scientific Clinical Centre of Pediatric Hematology, Oncology and Immunology named after Dmitry Rogache (Other)
Responsible Party: Sponsor
Other Study IDs: ASA-NIS-2023; NP (Other: Nizhpharm JSC)
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus Type 2; Coronary Artery Diseases; Aspirin Resistance
Keywords: chronic coronary syndrome; diabetes mellitus; platelet aggregation; resistance to acetylsalicylic acid
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients receiving the buffered form of ASA
- Group 2: Patients receiving the enteric-coated form of ASA

SUMMARY:
Patients with diabetes mellitus are characterized by "hyperreactive" platelets and a reduced response to ASA compared to individuals without diabetes. ASA that is absorbed in the intestine is slower to enter the bloodstream and become therapeutic concentrations compared to ASA that is absorbed in the stomach. It seems rational to test the hypothesis that the use of buffered ASA may be more effective in patients with diabetes and chronic coronary syndrome (CCS).

DETAILED DESCRIPTION:
Enteric-coated acetylsalicylic acid (ASA) is released more slowly and absorbed at lower concentrations over a longer period of time, which may result in lower ASA bioavailability and reduced antiplatelet effect compared to buffered ASA. Patients with diabetes mellitus are characterized by increased platelet reactivity and reduced pharmacodynamic response to ASA compared to nondiabetic individuals. It seems rational to test the hypothesis that administration of buffered ASA could be more effective in patients with diabetes and chronic coronary syndrome (CCS).

The first step to test this hypothesis (administration of buffered ASA could be more effective in patients with diabetes and chronic coronary syndrome (CCS)) was to conduct an observational study to detect ASA resistance in patients already receiving a buffered or enteric-coated form of ASA.

Rationale and background. Low doses of acetylsalicylic acid (ASA) are effective for the prevention of thrombotic events [1]. ASA inhibits platelet aggregation by irreversible acetylation and inactivation of the enzyme cyclooxygenase (COX). This prevents platelets and endothelium from converting arachidonic acid into prostaglandins and platelet-activating thromboxane (TX) [2]. ASA is known to cause gastrointestinal side effects, primarily dyspepsia or peptic ulcer disease [3]. Intestine-soluble coated forms of ASA have been developed to inhibit the breakdown of the drug in the stomach by releasing ASA in the proximal small intestine, suggesting that this may reduce the harmful effects of ASA on the gastric mucosa. Since enteric-coated ASA has been shown to cause significantly fewer minor asymptomatic gastrointestinal lesions compared to plain ASA as measured by endoscopy after short-term treatment [4]. However, the existing evidence that a truly enteric-coated ASA reduces gastrointestinal side effects such as resulting dyspepsia [5-7] or gastrointestinal bleeding of clinical significance [8] is questionable. This confirms that exposures severe enough to cause bleeding occur due to systemic rather than local effects of ASA [9]. However, there is a small amount of evidence that enteric coating may have adverse effects on the bioavailability and antiplatelet effects of ASA, especially in certain patient groups. Deacetylation of ASA to inactive salicylic acid occurs in the intestine and liver, the effect of the first passage through the liver (presystemic metabolism) is quite high, while the effect of the first passage through the small intestinal mucosa has not been determined [10]. ASA in the enteric soluble form is released more slowly and absorbed at lower concentrations for a longer period of time, which may result in lower ASA bioavailability and reduced antiplatelet effect compared to ASA in the plain form [11]. In the study by Cox et al. [12] with a crossover design studied 3 strategies: ASA in enteric soluble form 75 mg, ASA in plain form 75 mg, and the combination of dipyridamole 200 mg with ASA in plain form 25 mg (the combination was administered twice daily). Seventy-one healthy volunteers aged 20-50 years participated in the study. COX activity was measured in all before treatment and after 2 weeks of treatment. After a 2 week washout period, the study was repeated with a new drug for each study participant. The primary endpoint was inhibition of thromboxane A2 (TXA2) after 2 weeks of treatment. Treatment failure, defined as TXA2 inhibition less than 95%, was found in 0% [95% confidence interval (CI) 0-13.3%] of patients receiving ASA in plain form, 13% (95% CI 7.8-21.0%) in the group of patients with ASA in enteric soluble form, and 8% (95% CI 1.9-27.7%) in the combination treatment group. The study team concluded from these data that patients who take low-dose ASA preparations in enteric soluble form are less likely to receive the full benefit of ASA. In a study by Peace et al. [13] compared the effect of ASA in plain form and ASA in enteric soluble form on serum thromboxane B2 (TXB2) levels in patients with cardiovascular disease. Patients had been treated with ASA for at least 3 months and necessarily within 36 hours before the test. In 44 of 236 (19%) individuals, TXB2 levels were too high (>10 ng/mL), indicating an insufficient antiplatelet effect. To rule out pill noncompliance, 20 patients with elevated TXB2 levels took the pills under observation. Afterward, 10 patients still had TXB2 levels that were too high. All of these patients were receiving ASA in the enteric soluble form of 75 mg. These patients were changed to ASA in plain form at a dose of 75 mg and after 2 weeks of treatment, 7 of 10 (70%) had an adequate response (low TXB2 level). The three patients in whom an inadequate effect of ASA remained had an average weight of 120 kg, and after the dose was increased to 150 mg ASA in simple form, all three had an adequate reduction in COX activity. The authors concluded that the antiplatelet effect of ASA in the enteric soluble form may be insufficient even after multiple regular doses. This may be due to worse absorption, as most patients had a sufficient response to taking ASA in plain form. In addition, the results of the study showed that higher doses of ASA may be required in obese patients due to increased volume of distribution. Maree et al. [14] studied 131 stable patients with cardiovascular disease who received ASA in an enteric soluble shell at a dose of 75 mg. Elevated COX activity (TXB2>2.2 ng/mL) was found in 58 of 131 (44%) as a sign of inadequate antiplatelet effect. The authors found that inadequate reduction in COX activity was significantly associated with young age, high weight, and previous myocardial infarction. Thus, enteric coating may reduce the antiplatelet effect of ASA, which carries a risk of inadequate antithrombotic prophylaxis. Patients with DM2 are characterized by increased platelet reactivity and reduced pharmacodynamic response to aspirin compared to nondiabetic individuals [15,16]. This has been attributed to multiple mechanisms that are involved in the different profiles of pharmacodynamic response to antiplatelet therapy in DM2 patients. Among them, shortened lifespan and increased platelet turnover rate in patients with DM2, resulting in enhanced platelet regeneration, are thought to play an important role. Various approaches have been attempted to address the problem of aspirin resistance in a group of patients with CAD and DM2, there have been small studies with a change in dosing regimen with encouraging results, but there have been no large randomized trials that could change the current practice. And also considering the expert opinion [17] that the use of ASA in enteric soluble form is significantly safer than ASA in plain form in relation to the number of bleeding events is not supported by high levels of evidence, patients with reduced bioavailability of the drug (namely, people with a BMI greater than 35 kg/m2 or weight greater than 120 kg) should prefer ASA in plain form. From this statement, it seems rational to test the hypothesis that ASA should preferably be administered in a non-intestinal soluble form to patients in the DM and stable CHD group, who may also have reduced bioavailability to ASA. Most often, determination of COX activity (metabolites of TCA2 - TCEB2 in serum or 11-dehydrothromboxane B2 in urine) is used to confirm resistance to ASA, in the study of Gurbel [18] showed a non-linear relationship between serum TCEB2 inhibition and aggregometry. Aggregometry was null when TХB2 inhibition reached > 49%. Furthermore, the authors concluded: these results suggest that defining serum TХB2 inhibition > 95% to indicate the level of platelet COX-1 inhibition required to assess clinical efficacy may be overestimated and this should be reconsidered in future translational studies that attempt to relate ASA clinical efficacy to a threshold of laboratory measurements. Thus it is most appropriate to use aggregometry to assess clinical efficacy, which is what is planned to be performed in this study.

Sample size calculation. There are no studies assessing acetylsalicylic acid resistance when enteric-coated and buffered forms of acetylsalicylic acid are administered in patients with chronic coronary syndrome and type 2 diabetes mellitus. Therefore, the sample size calculation was based on the work published by Rocca et al. [19], in which the efficacy of different regimens and doses of acetylsalicylic acid in enteric-coated formulations on thromboxane A2 levels was evaluated in patients with diabetes mellitus through the assessment of its metabolites: serum thromboxane B2, 11-dehydrothromboxane B2 in urine. Taking into account that the evaluation of thromboxane A2 metabolites is a parameter by which the presence of resistance to acetylsalicylic acid is assessed, to some extent similar to the values of aggregometry according to the VerifyNow ASA test and correlating with it, it was assumed that it was possible to use the values of resistance to acetylsalicylic acid therapy according to the determination of thromboxane A2 metabolites to calculate the sample of our study. Thus, with 80% power at a two-sided significance level of 5% (α = 0.05), we needed to recruit 82 patients in each group to detect similar differences. Given the possible attrition of 20% of patients during the study, we planned to recruit 200 patients (100 patients in each group).

ELIGIBILITY:
Inclusion Criteria:

* Patients (men and women) aged 18 years and older with chronic coronary syndrome and DM2;
* Patient is taking Cardiomagnil (75 mg/day) - buffered form ASA or Aspirin® Cardio (100 mg/day) or Thrombo ACC® (100 mg/day) enteric-coated form ASA on a regular basis;
* Signed informed consent.

Exclusion Criteria:

* Patients with conditions that require anticoagulant therapy (e.g., atrial fibrillation, mechanical heart valves, etc.) or dual antiplatelet therapy (recent percutaneous coronary intervention, coronary bypass, myocardial infarction, cerebral infarction, etc.);
* Patients with severe renal disease (serum creatinine>2.5 mg/dL [221 micromol/L]) or estimated creatinine clearance <30 mL/min;
* Patients with a history of intracranial haemorrhage;
* Patients with any contraindications to acetylsalicylic acid, including known allergy or hypersensitivity to acetylsalicylic acid, drug excipients, or other nonsteroidal anti-inflammatory drugs;
* Patients with bronchial asthma induced by taking salicylates and non-steroidal anti-inflammatory drugs;
* Patients with erosive-ulcerous lesions of the gastrointestinal tract (in the exacerbation phase);
* Patients with future planned coronary bypass surgery, percutaneous coronary intervention or any other revascularisation in which dual antiplatelet therapy should be administered;
* Pregnant, lactating women;
* Patients with ongoing haemorrhage;
* Patients with known coagulopathies, thrombocytopathies, thrombocytopenia;
* Patients with active psychiatric, infectious diseases and cancer;
* Patients with chronic heart failure of New York Heart Association (NYHA) functional class III-IV (FC);
* Patients with congenital lactase deficiency, lactose intolerance, glucose-galactose malabsorption;
* Patients taking methotrexate (more than 15 mg per week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 adult patients of both sexes with an established diagnosis of CCS and DM2 who were prescribed buffered acetylsalicylic acid (Cardiomagnil) or acetylsalicylic acid in an enteric-coated form (Aspirin® Cardio or Thrombo ACC®) prior to inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Frequency of resistance to acetylsalicylic acid by VerifyNow Aspirin test | Evaluated one time. Patient has been taking acetylsalicylic acid in one of the forms with control of compliance for 7 preceding days before the test.
  Frequency of development of high residual platelet reactivity while taking acetylsalicylic acid in buffered form (Cardiomagnil) compared to taking acetylsalicylic acid in an enteric-coated form (Aspirin® Cardio/Trombo Ass®) according to the VerifyNow Aspirin clinical test.

SECONDARY OUTCOMES:
Frequency of acetylsalicylic acid resistance according to light transmission aggregometry results | Evaluated one time. Patient has been taking acetylsalicylic acid in one of the forms with control of compliance for 7 preceding days before the test.
  Frequency of development acetylsalicylic acid resistance while taking acetylsalicylic acid in buffered form (Cardiomagnil) compared to taking acetylsalicylic acid in an enteric-coated form (Aspirin® Cardio/Trombo Ass®) according to light transmission aggregometry results.
Combined clinical endpoint (any bleeding + re-hospitalisation for any cause + death) | Identified by call 180 days after inclusion in the study

CONTACTS AND LOCATIONS:
Overall Officials: Imad Akhmad Merai, Head of CCU, Study Chair — University Clinical Hospital na V.V.Vinogradov (branch of RUDN university na Patrice Lumumba)
Locations (1):
- University Clinical Hospital na V.V.Vinogradov (branch of RUDN university na Patrice Lumumba), Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Database, instrument data - aggregometry graphs.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Supporting information will be available after the publication of the article and indefinitely.
Access Criteria: Any researcher can get access, you just need to write to the contact email address